CLINICAL TRIAL: NCT01077427
Title: A Randomized Two-armed Open Study on the Adjuvant Therapy in Patients With R0/R1 Resected Pancreatic Carcinoma With Gemcitabine Plus Capecitabine (Arm GC) vs. Gemcitabine Plus Cisplatin With Regional Hyperthermia (Arm GPH)
Brief Title: Hyperthermia European Adjuvant Trial
Acronym: HEAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Collaborators: The European Society for Hyperthermic Oncology (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Rolf D. Issels, MD, PhD, Klinikum der Universitaet Muenchen, Grosshadern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115-09; 2008-004802-14 (EudraCT Number); AIO-PAK-0111 (Other: Arbeitsgemeinschaft Internistische Onkologie (AIO))
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Resected Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; adjuvant treatment; hyperthermia
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperthermia | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + Capecitabine (Active Comparator)
  Interventions: Drug: Gemcitabine + Capecitabine
- Gemcitabine + Cisplatin + regional hyperthermia (Experimental)
  Interventions: Device: Gemcitabine + Cisplatin + regional hyperthermia

INTERVENTIONS:
Device: Gemcitabine + Cisplatin + regional hyperthermia — Gemcitabine: 1000 mg/m² as iv-infusion on days 1 and 15 of each course (Total dose: 12 g/m²)
  Cisplatin: 25 mg/m² as iv-infusion on days 2, 3* and 16, 17* of each course (Total dose: 600 mg/m²)
  Regional hyperthermia: 60 minutes on days 2, 3*, and 16, 17* of each course
  * as an exception for medical or logistic reasons RHT and cisplatin can be applied day 4 instead of 3 and day 18 instead of 17
  Arms: Gemcitabine + Cisplatin + regional hyperthermia
Drug: Gemcitabine + Capecitabine — Gemcitabine: 1000 mg/m² as iv-infusion on days 1, 8 and 15 of each course (Total dose: 18 g/m²)
  Capecitabine: daily dose of 1660 mg/m²; administered orally for 21 days followed by 7 days' rest (one cycle) for six cycles
  Arms: Gemcitabine + Capecitabine

SUMMARY:
Improvement of the clinical outcome in patients with resectable pancreatic carcinoma through an intensified adjuvant treatment with gemcitabine, cisplatin and regional deep hyperthermia as compared to standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Any ductal adenocarcinoma of the pancreas confirmed by histology
2. Previous R0 or R1 resection of pancreatic tumor with a standardized procedure
3. No other previous or concomitant treatment of pancreatic carcinoma like radiation, neoadjuvant therapy or immunotherapy
4. No tumor recurrence after surgery
5. Performance status ECOG 0-2
6. Adequate bone marrow function defined as

   * WBC count ≥ 3.5 x 109/L and
   * platelets ≥ 150 x 109/L and
   * haemoglobin ≥ 9 g/dl documented within 1 week prior to randomization
7. Adequate renal function defined as

   * serum creatinine ≤ 1.2 mg/dL and
   * calculated GFR ≥ 60 mL/min documented within 1 week prior to randomization
8. Adequate coagulatory function defined as

   * Quick-value ≥ 70% and
   * aPTT ≤ 1.5 x ULN documented within 1 week prior to randomization
9. Transaminases (AST, ALT) ≤ 3 x ULN and bilirubin ≤ 2 x ULN documented within 1 week prior to randomization
10. At least 18 years of age
11. Women with childbearing potential and fertile men must use adequate contraceptive measures during and for at least 3 months (female) and 6 months (male) after completion of study therapy (Adequate methods for women are oral contraceptives with estrogen and progesterone, vaginal rings, contraceptive patches, estrogen-free ovulation inhibitors, intrauterine devices with progesterone, 3-month injections with depot progesterone, implants setting free progesterone, abstinence or sterilization (vasectomy) of the male partner. Men must use condoms.)
12. Women with childbearing potential must have a negative pregnancy test within 1 week prior to randomization (postmenopausal women with amenorrhea for more than 1 year are regarded as having no childbearing potential)
13. Written informed consent

Exclusion criteria:

1. Cystic carcinoma of the pancreas
2. Periampullary, papillary cancer
3. Metastatic disease
4. Presence of an active infection grade 3 or higher
5. Other severe disease which could impair the patient's ability to participate in the study according to the investigator's opinion
6. Pregnant or breastfeeding women
7. Known allergies or contraindications with regard to substances or procedures of study therapy
8. Severe, non-healing wounds, ulcers or bone fractures
9. Participation in another clinical trial during this study or within 4 weeks prior to randomization (Exception: participation in a surgical trial prior to this study, for instance RECOPANC trial, comparing two different surgical procedures of pancreas resection)
10. Past or current abuse of illegal or legal drugs or alcohol
11. Other primary malignant diseases in the medical history during the last 5 years (exceptions: carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin).
12. Permanent cardiac pacemaker
13. Clinically significant cardiovascular or vascular disease or disorder ≤ 6 months before study enrolment (e.g. myocardial infarction, unstable angina pectoris, chronic heart failure NYHA ≥ grade 2, uncontrolled arrhythmia, cerebral infarction
14. Gross adiposity defined as BMI > 40 kg/m²
15. Treatment with regional hyperthermia not possible for technical reasons (e.g. metal implant)
16. "Known documented dihydropyrimidine dehydrogenase (DPD) deficiency"

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause assessed up to 60 months

OTHER OUTCOMES:
Toxicity | Permanent assessment
Quality of Life | Permanent assessment
  EORTC QLQ C30

CONTACTS AND LOCATIONS:
Overall Officials: Rolf D. Issels, MD, PhD, Principal Investigator — Klinikum Grosshadern, Medical Center, University of Munich, Germany
Locations (1):
- Klinikum Grosshadern, Medical Center, University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Issels RD, Boeck S, Pelzer U, Mansmann U, Ghadjar P, Lindner LH, Albertsmeier M, Angele MK, Schmidt M, Xu Y, Bahra M, Pratschke J, Schoenberg M, Thasler WE, Salat C, Stoetzer OJ, Knoefel WT, Graf D, Wessalowski R, Keitel-Anselmino V, Koenigsrainer A, Bitzer M, Zips D, Bamberg M, Fietkau R, Ott O, Kawecki M, Wyrwicz L, Rutkowski P, Rentsch M, Ababei J, Reichardt P, Rigamonti M, Weber B, Abdel-Rahman S, Tschoep-Lechner K, Jauch KW, Bruns CJ, Oettle H, von Bergwelt-Baildon M, Heinemann V, Werner J; European Society for Hyperthermic Oncology (ESHO) and the German Arbeitsgemeinschaft Internistische Onkologie (AIO) Study Group for Pancreatic Cancer. Regional hyperthermia with cisplatin added to gemcitabine versus gemcitabine in patients with resected pancreatic ductal adenocarcinoma: The HEAT randomised clinical trial. Eur J Cancer. 2023 Mar;181:155-165. doi: 10.1016/j.ejca.2022.12.009. Epub 2022 Dec 30. PMID 36657324
- See also: Pankreaszentrum München — http://www.pankreaszentrum-muenchen.de